CLINICAL TRIAL: NCT03511911
Title: The Evaluation of Pelvic Floor Muscle Function: A Reliability and Correlation Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: JS-1548
Record Dates: First submitted 2018-04-13; First posted 2018-04-30 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-04

CONDITIONS: Pelvic Floor Dysfunction
Keywords: Pelvic floor muscle strength; modified Oxford Grading Scale; Levator ani testing; vaginal contraction pressure; reliability

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- GROUP A1 (Experimental): In GROUP A1, participants are all healthy women.A gynecological physician evaluates the participant's pelvic floor muscle strength by vaginal palpation based on modified Oxford Grading Scale(MOS) and Levator ani testing(LAT) without telling the participant her result, and records it on a unique paper other than in the Case Report Form.Then inspector A will test them twice using the PHENIX instrument with a 5 minutes' interval at the same day.After three days,participants in group A1 will be tested by inspector B twice in the same way as what they have done the first day.
  Interventions: Diagnostic Test: evaluation of pelvic floor muscle function through the PHENIX instrument; Diagnostic Test: vaginal palpation
- GROUP A2 (Experimental): In GROUP A2,participants are all healthy women.A gynecological physician evaluates participant's pelvic floor muscle strength by vaginal palpation without telling the participant her result, and records it on a unique paper other than in the Case Report Form as what GROUP A1 do.Then it is inspector B who will test them twice using the PHENIX instrument with a 5 minutes' interval at the same day.Three days later,participants in group A2 will be tested by inspector A twice in the same way as what they have done the first day.
  Interventions: Diagnostic Test: evaluation of pelvic floor muscle function through the PHENIX instrument; Diagnostic Test: vaginal palpation
- GROUP B1 (Experimental): In GROUP B1,patients are all with pelvic floor disorders.A gynecological physician evaluates the patient's pelvic floor muscle strength by vaginal palpation based on modified Oxford Grading Scale(MOS) and Levator ani testing(LAT) without telling the patient her result, and records it on a unique paper other than in the Case Report Form.Then inspector A will test them twice using the PHENIX instrument with a 5 minutes' interval at the same day.After three days,patients in group B1 will be tested by inspector B twice in the same way as what they have done the first day.
  Interventions: Diagnostic Test: evaluation of pelvic floor muscle function through the PHENIX instrument; Diagnostic Test: vaginal palpation
- GROUP B2 (Experimental): In GROUP B2,patients are all with pelvic floor disorders.A gynecological physician evaluates the patient's pelvic floor muscle strength by vaginal palpation without telling patient her result, and records it on a unique paper other than in the Case Report Form as what GROUP B1 do.Then it is inspector B who will test them twice using the PHENIX instrument with a 5 minutes' interval at the same day.Three days later,patients in group B2 will be tested by inspector A twice in the same way as what they have done the first day.
  Interventions: Diagnostic Test: evaluation of pelvic floor muscle function through the PHENIX instrument; Diagnostic Test: vaginal palpation
- GROUP C1 (Experimental): In GROUP C1,participants are all female who give birth to a child within a year(compliance and twice assessment are guaranteed,but PFMT are not allowed during the interval).A gynecological physician evaluates the participant's pelvic floor muscle strength by vaginal palpation based on modified Oxford Grading Scale(MOS) and Levator ani testing(LAT) without telling the participant her result, and records it on a unique paper other than in the Case Report Form.Then inspector A will test them twice using the PHENIX instrument with a 5 minutes' interval at the same day.After three days,participants in group C1 will be tested by inspector B twice in the same way as what they have done the first day.
  Interventions: Diagnostic Test: evaluation of pelvic floor muscle function through the PHENIX instrument; Diagnostic Test: vaginal palpation
- GROUP C2 (Experimental): In GROUP C2,participants are all female who give birth to a child within a year(compliance and twice assessment are guaranteed,but PFMT are not allowed during the interval).A gynecological physician evaluates the participant's pelvic floor muscle strength by vaginal palpation without telling patient her result, and records it on a unique paper other than in the Case Report Form as what GROUP C1 do.Then it is inspector B who will test them twice using the PHENIX instrument with a 5 minutes' interval at the same day.Three days later,participants in group C2 will be tested by inspector A twice in the same way as what they have done the first day.
  Interventions: Diagnostic Test: evaluation of pelvic floor muscle function through the PHENIX instrument; Diagnostic Test: vaginal palpation

INTERVENTIONS:
Diagnostic Test: evaluation of pelvic floor muscle function through the PHENIX instrument — the PHENIX instrument was designed and produced for sensing muscle activity with surface electrodes, pressure probes and external captors,so it could test biological signals of pelvic floor muscle in human body.
Diagnostic Test: vaginal palpation — vaginal palpation is based on modified Oxford Grading Scale(MOS) and Levator ani testing(LAT) to test patients' pelvic muscle strength

SUMMARY:
1. To explore the correlations among measures of PFM strength between using vaginal palpation quantified by modified Oxford Grading Scale and Levator ani testing and manometry in PHENIX instrument;
2. To determine the intra- and inter-rater reliability of PFM strength measured using manometry in PHENIX instrument.

DETAILED DESCRIPTION:
This is a study using a randomized crossover blind method.All the volunteers are divided into 2 groups randomly. At the first time, a gynecological physician evaluates patient's pelvic floor muscle strength by vaginal palpation based on modified Oxford Grading Scale(MOS) and Levator ani testing(LAT) without telling patient her result, and record it on a unique paper other than in the Case Report Form.

At the same day, patient will be tested by inspector A or B randomly twice with the PHENIX instrument.A 5 minutes' interval is needed between two tests in order to reduce the possibility of fatigue of pelvic floor muscles. The outcome is secretive to the patient as well.

A second time evaluation is required in 3 days' later by a different inspector from the first time.(interrater and intrarater) All the data including strength of MOS and LAT, the outcomes by inspector A and B, cannot be collected together and told to the patient until she finished the whole process.

Pelvic floor muscle training is not permitted during the evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. Having sex life and tolerable to vaginal examination
2. Planning to live locally for a long time

Volunteers are divided into three groups Group A: healthy women

1. healthy women for physical examination
2. except in the first year after delivery,duration of lactation or with a clear diagnosis as pelvic organ prolapse beyond the level of hymen or incontinence.

Group B:patients with pelvic floor disorders

1. patients diagnosed as incontinence by clinical presentation(patients with urinary incontinence are required to complete the questionnaire of ICIQ-SF)
2. patients with pelvic organ prolapse beyond the level of hymen
3. except in the first year after delivery,duration of lactation and patients with chronic pelvic pain

Group C: female who give birth to a child within a year(compliance and twice assessment are guaranteed,but PFMT are not allowed during the interval)

Exclusion Criteria:

1. Patients who are undergoing pelvic floor muscle training
2. History of radical operation of pelvic cavity(cervical cancer,rectal cancer,bladder cancer, ect）
3. History of pelvic radiotherapy
4. History of pelvic floor surgery
5. Duration of pregnancy
6. Latex allergy
7. Colpitis
8. Operation on pelvis within 6 months

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2018-06-11 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum vaginal contraction pressure | 3 days
  Maximum vaginal contraction pressure is evaluated by manometry

SECONDARY OUTCOMES:
vaginal rest pressure | 3 days
  measure when no vaginal contraction by manometry
Pelvic floor muscle strength | 1 day
  The modified Oxford Grading Scale is used to quantify PFM strength through vaginal palpation
Pelvic floor muscle strength（repitition） | 1 day
  Levator ani testing is used to quantify PFM strength
Pelvic floor muscle contraction endurance | 3 days
  muscle contractions maintained for 0 s are defined as grade 0,and 5 s or longer as grade V. Normal muscles can maintain the contraction for 5 s. The endurance is measured by PHENIX instrument.
pelvic organ prolapse quantification(POP-Q) | 1 day
  POP-Q is measured when maximum valsalva

CONTACTS AND LOCATIONS:
Overall Officials: Lan Zhu, MD, Principal Investigator — Peking Union Medical College Hospital, Chinese Academy of Medicine Sciences
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medicine Sciences, Beijing, Beiing, China